CLINICAL TRIAL: NCT01083407
Title: Oral Care Interventions With 0.12% Chlorhexidine and Ventilator Associated Pneumonia in Critically Ill Children: Prospective, Randomic and Double Blind Study
Brief Title: Oral Care Interventions and Ventilator Associated Pneumonia in Critically Ill Children
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Federal University of São Paulo (Other)
Collaborators: Fundação de Amparo à Pesquisa do Estado de São Paulo (Other Government)
Responsible Party: Federal University of São Paulo, Nursing Department
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: Oral care and VAP in children.
Record Dates: First submitted 2010-03-05; First posted 2010-03-09 (Estimated); Last update posted 2010-03-09 (Estimated); Status verified 2009-03

CONDITIONS: Ventilator Associated Pneumonia
Keywords: Oral care.; Chlorhexidine.; Pediatric Nursing; Intensive Care; Nosocomial infection; Pneumonia; Oropharyngeal colonization; Tracheal colonization
MeSH Terms: conditions — Pneumonia, Ventilator-Associated; Cross Infection; Pneumonia | interventions — chlorhexidine gluconate; Toothbrushing

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 0.12% Chlorhexidie Digluconate (Experimental): Oral care included use of an oral gel containing chlorhexidine digluconate 0.12% as an active ingredient (chlorhexidine digluconate 0.12%; methylcellulose gel 2.12%, 25 g; gooseberry syrup, 4 drops; menthol solution 50%,3 drops; and distilled water, to 30 g).The gel is applied on a toothbrush, and the teeth are cleaned in quadrants; all teeth surfaces are cleaned (vestibular,lingual, occlusal, and incisal). After each quadrant was cleaned, 10 mL of water (dispensed via a syringe) is used to rinse the quadrant and continual aspiration is used to remove all the gel and debris. After all the teeth are cleaned, the ventral surface of the tongue is brushed with posteriorto- anterior movements.
  Interventions: Drug: 0.12% Chlorhexidine Digluconate
- Toothbrushing (Placebo Comparator): This group received the same oral care that experimental group with the use of a similarly formulated gel without the antiseptic agent.The gel is applied on a toothbrush, and the teeth are cleaned in quadrants; all teeth surfaces are cleaned (vestibular, lingual, occlusal, and incisal). After each quadrant is cleaned, 10 mL of water (dispensed via a syringe) is used to rinse the quadrant and continual aspiration is used to remove all the gel and debris. After all the teeth are cleaned, the ventral surface of the tongue is brushed with posteriorto-anterior movements.
  Interventions: Other: Toothbrushing

INTERVENTIONS:
Drug: 0.12% Chlorhexidine Digluconate — Oral care with 0.12% Chlorhexidine Digluconate and toothbrushing is realized twice a day and took about 10 minutes to complete, depending on the child's acceptance and clinical conditions.
  Arms: 0.12% Chlorhexidie Digluconate
Other: Toothbrushing — Gel is applied on a toothbrush, and the teeth are cleaned in quadrants; all teeth surfaces are cleaned (vestibular, lingual, occlusal, and incisal). After each quadrant is cleaned, 10 mL of water (dispensed via a syringe) is used to rinse the quadrant and continual aspiration is used to remove all the gel and debris. After all the teeth are cleaned, the ventral surface of the tongue is brushed with posteriorto-anterior movements.
  Arms: Toothbrushing

SUMMARY:
This experimental study aims to verify the influence of the oral hygiene performance with chlorhexidine digluconate 0.12% in the development of VAP in children. The data collection begun in April, 2005 during the performance of the masters degree course dissertation entitled "Clinical study about the effect of the oral hygiene with chlorhexidine digluconate 0.12% in the oropharynx colonization of children in intensive care", being performed in a PICU of nine beds in a university hospital in the city of São Paulo, after approval of the Research Ethics Committee of the institution. The study is composed by three types of variables: Independent variable, dependent variables, and complementary variables. The categorical variables will be analyzed in accordance with the Person's Chi-Square test of or Fisher's exact test. The numerics will be submitted to the analysis of variance ANOVA or Kruskall Wallis. For variables with heterogeneous distribution between the groups, the multivariate analysis will be applied to the evaluation of the influence in the determination of the development risk of the dependent variable. The rejection level will be fixed in 0.05 of the nullity hypothesis.

DETAILED DESCRIPTION:
Recent progress in identification of oral microorganisms has shown that the oropharynx can be a site of origin for dissemination of pathogenic organisms to distant body sites, such as the lungs. THe aims of the study were to compare the oropharyngeal microbiological profile, VAP incidence, duration of mechanical ventilation, and length of stay in the intensive care unit of children receiving mechanical ventilation who had pharmacological or nonpharmacological oral care.

A randomized and controlled study has been performed in a pediatric intensive unit in São Paulo, Brazil. The children are randomly assigned to an experimental group that received oral care with use of 0.12% chlorhexidine digluconate or a control group that received oral care without an antiseptic. Oropharyngeal and tracheal secretions were collected and cultured on days 0, 2, and 4, and at discharge.

ELIGIBILITY:
Inclusion Criteria:

* Critically ill children.
* Age: 29 days to 18 years.

Exclusion Criteria:

* Newborn age.
* Pneumonia at PICU admission.
* Tracheostomy.
* Tracheal intubation higher than 24 hours in the PICU admission.
* PICU LOS lower than 48 hours.
* Responsibles declined consent.

Ages: 29 Days to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 146 (Actual)
Dates: Start 2005-06; Primary Completion 2006-06 (Actual); Study Completion 2008-06 (Actual)

PRIMARY OUTCOMES:
Ventilator associated pneumonia | 48 hours after tracheal intubation
  Influence of oral care with 0.12% chlorhexidine on VAP incidence diagnosed by clinical pulmonary infection score.

SECONDARY OUTCOMES:
PICU Lengh of Stay | Necessary days to PICU discharge
  Influence of oral care with 0.12% chlorhexidine on PICU LOS
Time of Mechanical pulmonary ventilation | Last day of MPV
  Influence of oral care with 0.12% chlorhexidine on time of mechanical ventilation.

REFERENCES:
- [Derived] Kusahara DM, Friedlander LT, Peterlini MA, Pedreira ML. Oral care and oropharyngeal and tracheal colonization by Gram-negative pathogens in children. Nurs Crit Care. 2012 May-Jun;17(3):115-22. doi: 10.1111/j.1478-5153.2012.00494.x. Epub 2012 Feb 23. PMID 22497915